CLINICAL TRIAL: NCT03379961
Title: Identification of Social Categorisation Process Who Intervene During Patient Nurse Triage and Research of Them Impacts in Cares.
Brief Title: Identification and Research of Impacts of Social Categorization Process in Nurse Triage (SOCIAL SORTING)
Acronym: SOCIALSORTING
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRIP-16-0206
Record Dates: First submitted 2017-12-07; First posted 2017-12-20 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Socialised Disturbance of Conduct
Keywords: social categorization; nurse sorting; emergencies units

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Social Sorting is a: non interventional, observational, qualitative and multicenter research. It investigates three French emergency units in three French centers (UH of Angers, H of Le Mans, H of Laval).

It is a research based on nursing sciences and social-psychology and it proposes to study the process of social categorization that intervenes during triage nursing.

The process of social categorization has developped since the beginning of XX century (LIPPMANN, in 1922, in United States, he gave the first definition of stereotype// DURKHEIM, in France described step by step the individuals and the collectives representations.

During XX century the social psychology developed a lot of studs about group dynamics (social categorization, influence phenomenon, conspiracy theories,...) within several domains : industry, politics, public services as police, social units,... and also in healthcare (but always about a social categorisation in particular and often with a limited study of impacts).

Social Sorting includes all social categorization as possible and search to do a scientific evaluation of their impact.

DETAILED DESCRIPTION:
Emergencies units are a special way to access at cares. These units must continually adapt their practice because it is impossible to predict patient's flow, number of hospital's available beds and kinds of emergencies (medical, chirurgical, psychiatric, social). Organization and quality of cares are based on a balance between competences and human attributes.

The first step in medical care takes place thanks to the nurse triage. They must summarize a lot of information about patients ( such as medical letters, firemen's transmission,...) and make a quick clinical exam. This action permits to determine an emergency degree and prioritize it. This activity is based on clinical categorization and clinical tools (scales of triage).

The clinical categorization is a professional competence (nurses learn what categorization is at school and develop it at hospital).In this research social categorization will be confronted with another type of categorization : the social categorization.

The latter it is very different categorization, in fact, it is shared by anybody (nonprofessionals of healthcare and professionals). The social categorization can be described like the phenomenon that permits to simplify the reading of the world. That also permits for anybody to define itself and define the one or more group membership. That process is continually in movement (social prejudices changes according to History, depending on the place of the world htat person lives,...).

The social categorization process has a real impact on action, thinking and relation with the world and the others persons.

The social categorization reveals its process in prejudice (sensitive dimension), stereotypes(cognitive dimension, stereotypes are organized around a central trait and others peripherals traits) and conducts to discrimination (behavior dimension) about origins, diseases, age,....Social categorization provides of naive theorization about social objects. For instance, a man who stereotypes woman with blond hair thinking "she is stupid" when he sees her in the street ( that it is a prejudice, a central trait) and this feeling conducts him to think "she is superficial, she does not work, she watches reality TV show everyday,..."(that it is a stereotype with peripherals traits). If this same man does not accept to help this woman if she needs him, it can considered like discrimination.

A lot of studies in public administrations have shown the important influence of social categorization on power which exists in any relations and the non-personalization as final response. In healthcare domain for instance, the research of WILLIAMS have shown existence of "bads patients".

Our first hypothesis is that process of social categorization exists and it has several faces(potentially negative). We also make the hypothesis that they have impacts on several aspects of medical care like : waiting time, management of pain,....We finally do the hypothesis that exist links between : the presence of process of social categorization in triage nursing and : individual traits (race, sex, age,...), specificities of any contexts.

Social Sorting wishes to identify with scientific measure the presence of social categorization process in triage nursing and it is unprecedented.

Then it is also to describe the impacts of this process on several parts of the medical care.

It could be interesting to improve nursing staff. It could be also interesting to patients because it is the equality of health offer which is asked in Social Sorting. In France, in 2015, 10 billions of patients came in emergency units. The study of feasibility wich was done before Social Sorting has shown that 20 percent of nurses sorting include social categorization nurse.

The results of this research could interest professional of healthcare domain and socio-psychologist.

ELIGIBILITY:
Inclusion Criteria:

* all nurses who accept micro and all patients over the age of majority

Exclusion Criteria:

* all nurses who do not accept micro and all minor patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Investigators wish a participation equal or superior to 50 percent of total number of nurses in centers.
  504 triage nurses will be include, it represent 168 per center (one an hour during a week), 6 per periods (nights, days, weeks, weekends). We justify this choice by desire to produce qualitative and exhaustive results and necessity to respect constraints, practicability and cost.
Sampling Method: Probability Sample
Enrollment: 504 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-02-17 (Actual); Study Completion 2018-02-17 (Actual)

PRIMARY OUTCOMES:
Number of patient stigmatized during nurse triage | 5 months
  It is the percent of patient stigmatised among the 504 contexts of triage nursing observed. To determine that, each situation of triage nursing will be examined by three analysts individually. After this time of individual analysis, there will be a time of collegial analysis. To consider that a nurse triage include social categorization it will take a collegial decision-making. A patient is considered like stigmatized when one or several social traits are mentioned during it triage nursing. For instance, if a fireman brings with a patient with twisted ankle and if he mentions that a patient is homosexual during his transmission. Homosexuality in this situation has not interest to taking care. It would have been different if this same patient were come to treat a sexual infection.

SECONDARY OUTCOMES:
Nature of social categorization | 5 months
  the description of the social categorization process observed during the triage, its nature (including verbal, non-verbal and written categorization) and themes (sociocultural origin, sex, age...). To determine that, each situation of nurse triage will be examined by three analysts individually. After this time of individual analysis, there will be a time of collegial analysis. For each analysis, analysts will have to define if one social categorization is mentions on verbal only or in non-verbal too for instance.
Risk factors of social categorization | 5 months
  The research of links between the social categorization process in triage nursing and the risk factors which may increase the presence of it. The factors examined are : the context of sorting (flow of patients, people who are presents during the triage...) the specificities of any players in care relationship (sex, age, behavior...), the level of aggressiveness ( does it have a link between the presence of a social categorization and the level of aggressiveness ?). To determine that, analysts will compare if, for example, all patients coming for abdominal pain (with same clinical exam, same level of pain) during a sunday night will be sort similarly.
Links between social categorisation and elements of medical care | 5 months
  the research of links between the existence of a social categorization process during the sorting and elements of medical care (waiting time, quality and nature of installation, pain support,...). To determine that analysts will compare if all patients, for example, wich coming with dyspnea (with same clinical exam) will be evaluate with the same emergency level or if subsaharan patients will be evaluate diferently.

CONTACTS AND LOCATIONS:
Overall Officials: Pilleron BP Benjamin, nurse, Principal Investigator — UH Angers
Locations (3):
- France (3):
  - CHU Angers, Angers
  - CH Laval, Laval
  - CH Le Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pilleron B, Douillet D, Furon Y, Haubertin C, Parot-Schinkel E, Vielle B, Roy PM, Poiroux L. Nurses' moral judgements during emergency department triage - A prospective mixed multicenter study. Int Emerg Nurs. 2024 Aug;75:101479. doi: 10.1016/j.ienj.2024.101479. Epub 2024 Jun 26. PMID 38936277